CLINICAL TRIAL: NCT06039293
Title: Program AACTIVE: African Americans Coming Together to Increase Vital Exercise
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study underwent some protocol re-design that prompted a new IRB, thus this study never commenced.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jaclynn Hawkins, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00234526
Record Dates: First submitted 2023-08-25; First posted 2023-09-15 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes; Depression
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive 10 cognitive behavioral therapy sessions and 6 physical activity sessions over 12 weeks. Participants in this group will also be assigned exercise goals. Exercise goals will be adapted to accommodate the physical and medical restrictions of older adults with type 2 diabetes. Exercise goals consistent with our prior trials will be used using a stepwise approach starting with 100 minutes of aerobic activity in week 1, 125 minutes in week 2 and 150 minutes in weeks 3 through 12. Exercise prescriptions will be based on the results obtained from the 6 Minute Walk Test obtained at baseline
  Interventions: Behavioral: Cognitive behavioral therapy and physical activity sessions
- Control (Other): Participants in the control group will receive enhanced usual care and will not take part in cognitive behavioral therapy sessions or exercise sessions. The EUC group will receive the American Diabetes Association "Diabetes Basics" web series (one video per week for 10 weeks) or "Diabetes Basics" handouts sent via mail.
  Interventions: Behavioral: Enhanced Usual Care + Diabetes Basics Web Series

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy and physical activity sessions — The intervention group will receive 10 sessions of cognitive behavioral therapy (CBT) and 6 physical activity sessions over the 12-week period. All Program AACTIVE CBT sessions and exercise sessions will run concurrently and take place virtually using Master of Social Work (MSW) trainees and Movement Science Master of Science students from the University of Michigan.
  Arms: Intervention
Behavioral: Enhanced Usual Care + Diabetes Basics Web Series — Participants will receive the American Diabetes Association "Diabetes Basics" web series (one video per week for 10 weeks) or "Diabetes Basics" handouts sent via mail.
  Arms: Control

SUMMARY:
Program AACTIVE will enroll 80 African American/Black men with type 2 diabetes and depression. Participants will be randomized to either the intervention arm or the control arm. Participants in the intervention arm will receive counseling (cognitive behavioral therapy) and physical activity sessions over 12 weeks. Counseling and physical activity sessions will take place via a video conferencing platform. There will also be 3 in-person health assessments including baseline, at 12-weeks and 3-month follow up. The investigators are interested in seeing if physical activity and counseling improve A1C outcomes and depression symptoms for participants.

DETAILED DESCRIPTION:
Participants will be randomized to the Program AACTIVE intervention group or an Enhanced Usual Care (EUC) group. The intervention group will receive 10 sessions of cognitive behavioral therapy (CBT) and 6 physical activity sessions over the 12-week period. All Program AACTIVE CBT sessions and exercise sessions will run concurrently and take place virtually.

ELIGIBILITY:
Inclusion Criteria:

* African American/Black males, ambulatory status, diagnosed with type 2 diabetes for one year duration or longer, PHQ-9 score >=15 with no self-reported psychotic symptoms, live in the Wayne or Washtenaw Counties, have reliable transportation to in-person events, have reliable access to internet and a device that supports video calls.

Exclusion Criteria:

* Stage 2 hypertension as defined by JNCVIII, recent cardiac events, recent laser surgery for proliferative retinopathy, history of stroke, lower limb amputation, peripheral neuropathy, aortic stenosis or other sever valvular heart disease, atrial fibrillation, severe COPD (e.g., basal oxygen), class III or IV heart failure or medical instability.

Participants who are currently receiving psychotherapy services for the treatment of depression from a mental health care provider will be excluded while participants who are currently receiving only medication management from as psychiatrist will be included.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1C % | baseline, 3-months (post intervention), 6-months (3-month follow up)
  Finger poke
Change in Depressive Symptoms | baseline, 3-months (post intervention), 6-months (3-month follow up)
  Patient Health Questionnaire-9 Scale, a scale to measure depression severity. Scores less than 5 almost always signified the absence of a depressive disorder; scores of 5 to 9 predominantly represented patients with either no depression or subthreshold (i.e., other) depression; scores of 10 to 14 represented a spectrum of patients; and scores of 15 or greater usually indicated major depression.
Blood Pressure | baseline, 3-months (post intervention), 6-months (3-month follow up)
  Digital Blood Pressure Machine measuring systolic and diastolic blood pressure. Blood pressures will be measured twice and averaged. The average will be recorded as the blood pressure reading.
Heart Rate | baseline, 3-months (post intervention), 6-months (3-month follow up)
  Digital Blood Pressure Machine (with heart rate measure)
Physical Activity Minutes Each Week | Weekly, for intervention period between baseline and 3 months (post intervention)
  Minutes of physical activity each week logged in a physical activity log.
Number of Steps | Weekly, for intervention period between baseline and 3 months (post intervention)
  Fitbit (provided by the study) readings and physical activity log

SECONDARY OUTCOMES:
Diabetes Quality of Life | baseline, 3-months (post intervention), 6-months (3-month follow up)
  The Diabetes Quality of Life Brief Clinical Inventory contains 15 items, with response options ranging from 1 ("Very Satisfied") to 5 ("Very Dissatisfied"). Possible scores range from 15 to 75. Lower scores suggest a satisfactory quality of life.
General Quality of Life | baseline, 3-months (post intervention), 6-months (3-month follow up)
  Short Form-12 Scale (SF-12). The 12 response options are coded as follows: 1=yes, limited a lot; 2=yes, limited a little; 3=no, not limited at all. A higher score is indicative of better health.

OTHER OUTCOMES:
Diabetes Self-Efficacy | baseline, 3-months (post intervention), 6-months (3-month follow up)
  Perceived Diabetes Self-Management Scale (PDSMS). The responses for the PDSMS items range from 1 = "Strongly Disagree" to 5 = "Strongly Agree." Four of the items (#s 1, 2, 6, & 7) are worded such that high agreement signifies low self-efficacy or perceived competence. These four items are reverse scored prior to being added to the other four items. The total PDSMS score can range from 8 to 40, with higher scores indicating more confidence in self-managing one's diabetes.
Masculinity Ideology | baseline, 3-months (post intervention), 6-months (3-month follow up)
  Conformity to Masculine Norms Inventory (CMNI-30). The 30-item scale contains 10 subscales (three items per subscale). Response options range from 0 ("strongly disagree") to 5 ("strongly agree"). Items within each subscale are averaged and then summed across all subscales. Higher scores represent stronger conformity to traditional masculine norms.
BMI | baseline, 3-months (post intervention), 6-months (3-month follow up)
  kilograms/meters squared
Social Support | baseline, 3-months (post intervention), 6-months (3-month follow up)
  Duke-UNC Functional Social Support Questionnaire. This is an 8 question scale and responses to each question are scored on a 1 to 5 scale. "As much as I would like" receives a score of 5 and "Much less than I would like" receives a score of 1. The scores from all eight questions are summed (maximum 40) and then divided by 8 to get an average score. The higher the average score, the greater the perceived social support.
Diabetes-related Distress | baseline, 3-months (post intervention), 6-months (3-month follow up)
  Type 2 Diabetes Distress Assessment System. The scale is comprised of an 8-item Core Tool, and a Sources Tool that examines seven distinct Sources of diabetes distress, each containing three items. On a 5-point Likert scale, response options range from 1 ("not a problem") to 5 ("very serious problem"). A higher Core diabetes distress score has been associated with higher HbA1c levels, BMI, and poorer self-management behaviors. There are no established thresholds for what would be considered "elevated" diabetes distress.
Prescribed Medication Adherence | baseline, 3-months (post intervention), 6-months (3-month follow up)
  Adherence to Refills and Medicines Scale for Diabetes (ARMS-D). ARMS-D is a 12-item scale with response options ranging from 1 ("none of the time") to 4 ("all of the time"). Scores are summed (range: 12 to 48), where higher scores are indicative of greater difficulty taking diabetes medications.
Aerobic Capacity | baseline, 3-months (post intervention), 6-months (3-month follow up)
  6 Minute Walking Test

CONTACTS AND LOCATIONS:
Overall Officials: Jaclynn Hawkins, PhD, Principal Investigator — University of Michigan, School of Social Work

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data with other researchers.